CLINICAL TRIAL: NCT00424528
Title: A Two-Week, Randomized, Modified-Blind, Double-Dummy, Parallel-Group Efficacy and Safety Study of Arformoterol Tartrate Inhalation Solution Twice-Daily, Tiotropium Once-Daily, and Arformoterol Tartrate Inhalation Solution Twice-Daily and Tiotropium Once Daily in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy Safety Study of Arformoterol/Tiotropium Combination Versus Either Therapy Alone in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 091-902
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2009-04-02 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Bronchitis; Emphysema
Keywords: COPD including chronic bronchitis and emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema | interventions — Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arformoterol 15 mcg twice daily (Active Comparator): Arformoterol 15 mcg twice daily/Placebo Inhalation Powder
  Interventions: Drug: Arformoterol Tartrate Inhalation Solution; Drug: Placebo
- Tiotropium 18 mcg once daily (Active Comparator): Tiotropium 18 mcg once daily/Placebo Inhalation Solution
  Interventions: Drug: Tiotropium; Drug: Placebo
- Arformoterol /Tiotropium (Experimental): Arformoterol 15 mcg twice daily/Tiotropium 18 mcg once daily
  Interventions: Drug: Arformoterol and Tiotropium

INTERVENTIONS:
Drug: Arformoterol Tartrate Inhalation Solution — Arformoterol tartrate inhalation solution 15 mcg twice daily and placebo inhalation powder once daily.
  Other Names: Brovana®
  Arms: Arformoterol 15 mcg twice daily
Drug: Tiotropium — Placebo inhalation solution twice daily and tiotropium inhalation powder 18 mcg once daily.
  Other Names: Spiriva
  Arms: Tiotropium 18 mcg once daily
Drug: Arformoterol and Tiotropium — Arformoterol tartrate inhalation solution 15 mcg twice daily and Tiotropium inhalation powder 18 mcg once daily.
  Other Names: Brovana; Spiriva
  Arms: Arformoterol /Tiotropium
Drug: Placebo — Placebo inhalation solution and placebo inhalation powder
  Arms: Arformoterol 15 mcg twice daily; Tiotropium 18 mcg once daily

SUMMARY:
The purpose of this study is to evaluate and compare the efficacy of arformoterol twice a day and tiotropium once a day (dosed sequentially) versus tiotropium once a day alone in subjects with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, modified-blind, double-dummy two-week parallel-group efficacy and safety study of arformoterol tartrate inhalation solution twice daily, tiotropium inhalation powder once daily and arformoterol tartrate inhalation solution twice daily and tiotropium inhalation powder once daily (dosed sequentially) in subjects with COPD. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be at least 45 years old at the time of consent.
* Subjects must have a pre-established primary clinical diagnosis of COPD.
* Subjects must have a baseline FEV1 of ≤65% of predicted normal value at Visit 1.
* Subjects must have a FEV1 ≥ 0.70L at Visit 1.

Exclusion Criteria:

* Subjects who do not have a FEV1/forced vital capacity (FVC) ratio of ≤70% at Visit 1.
* Subjects who do not have a ³15 pack-year smoking history and a baseline breathlessness severity grade of ³2 (Modified Medical Research Council [MMRC] Dyspnea Scale Score) at Visit 1.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Andrews, M.D., Study Director — Sumitomo Pharma America, Inc.
Locations (28):
- United States (28):
  - Jasper, Alabama
  - Tucson, Arizona
  - San Diego, California
  - Colorado Springs, Colorado
  - DeFuniak Springs, Florida
  - DeLand, Florida
  - Topeka, Kansas
  - Hazard, Kentucky
  - Madisonville, Kentucky
  - Marrero, Louisiana
  - Sunset, Louisiana
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Saint Charles, Missouri
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Eugene, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - East Providence, Rhode Island
  - Lincoln, Rhode Island
  - Columbia, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Knoxville, Tennessee
  - Tacoma, Washington
  - Morgantown, West Virginia

REFERENCES:
- [Derived] Tashkin DP, Donohue JF, Mahler DA, Huang H, Goodwin E, Schaefer K, Hanrahan JP, Andrews WT. Effects of arformoterol twice daily, tiotropium once daily, and their combination in patients with COPD. Respir Med. 2009 Apr;103(4):516-24. doi: 10.1016/j.rmed.2008.12.014. Epub 2009 Feb 8. PMID 19208459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter (34 sites) study.
Pre-assignment Details: Started: consists of all subjects who were randomized to treatment and received at least one dose of randomized study drug (Intent to treat population). One patient was randomized to the arformoterol/tiotropium group but discontinued before receiving any study medication and is therefore not included.
Period: Overall Study
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Started | 76 | 80 | 78
Completed | 71 | 76 | 74
Not Completed | 5 | 4 | 4
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — noncompliance with study requirements | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium | Total
Number analyzed (Participants) | 76 | 80 | 78 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 50 | 52 | 149
  >=65 years | 29 | 30 | 26 | 85
Age Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.4) | 61.2 (9.5) | 62.2 (7.6) | 61.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 36 | 110
  Male | 39 | 43 | 42 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 6 | 7 | 18
  White | 71 | 74 | 70 | 215
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 80 | 78 | 234
Number of Pack Years Smoked [Number; unit: Participants] — Number of participants with a particular range of pack years smoked.
  Participants
    >=15 years to <25 years | 0 | 1 | 6 | 7
    >=25 years to <=30 years | 4 | 4 | 4 | 12
    >=30 years | 72 | 75 | 68 | 215
Packs per day currently smoked [Number; unit: Participants] — Number of participants with a particular range of packs per day currently smoked.
  Participants
    >0 to 1 pack | 24 | 30 | 22 | 76
    >1 to 2 packs | 22 | 24 | 16 | 62
    >2 to 4 packs | 3 | 0 | 1 | 4
    >4 packs | 0 | 0 | 0 | 0
    Currently does not smoke | 27 | 26 | 39 | 92
Baseline Dyspnea Index (BDI) Focal Score [Mean (Standard Deviation); unit: units on a scale] — Baseline Dyspnea Index(range 0-12) is defined to be the sum of the Functional Impairment, Magnitude of Task, and Magnitude of Effort scores (each on a 0-4 scale) obtained at visit 2 (baseline. On each scale, a high measurement represents the most impairment to health.
  units on a scale | 5.8 (2.0) | 5.8 (1.9) | 5.5 (2.1) | 5.7 (2.0)
Best Forced Expiratory Volume in one second (FEV1)/Best Forced Vital Capacity (FVC) ratio [Mean (Standard Deviation); unit: Liters] | 0.510 (0.098) | 0.514 (0.107) | 0.525 (0.108) | 0.516 (0.104)
FEV1 [Mean (Standard Deviation); unit: Liters] | 1.366 (0.457) | 1.377 (0.460) | 1.350 (0.408) | 1.365 (0.440)
FEV1 Percent Predicted [Mean (Standard Deviation); unit: percent predicted of FEV1] | 45.4 (11.9) | 45.7 (11.5) | 44.9 (12.0) | 45.4 (11.8)
Inspiratory Capacity [Mean (Standard Deviation); unit: Liters] | 2.005 (0.615) | 1.979 (0.555) | 1.924 (0.516) | 1.969 (0.562)
Modified Medical Research Council Dyspnea Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Dyspnea scale score reflects the highest numbered question to which the subject answered "yes" in a series of five questions, each describing progressively worse dyspnea. Scores range from 0 to 4, with a score of 4 indicating that a subject is too breathless to leave the house or becomes breathless when dressing or undressing.
  units on a scale | 2.7 (0.6) | 2.9 (0.7) | 2.9 (0.6) | 2.8 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Time-normalized Area Under the Change From Study Baseline Curve for Forced Expiratory Volume in One Second (FEV1) Over 24 Hours (nAUC0-24B)
Time Frame: 24 hours following two weeks of dosing.
Population: Total number of subjects in each arm: 76, 80, 78
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 71 | 75 | 72
Liters | 0.104 [0.054 to 0.155] | 0.080 [0.035 to 0.124] | 0.221 [0.175 to 0.267]
Statistical Analysis 1: Comparison: Arformoterol 15 Mcg Twice Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA; Study baseline FEV1 as covariate and treatment group as fixed effect
Statistical Analysis 2: Comparison: Tiotropium 18 Mcg Once Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA; Study Baseline FEV1 as a covariate and treatment group as a fixed effect
Statistical Analysis 3: Comparison: Arformoterol 15 Mcg Twice Daily vs Tiotropium 18 Mcg Once Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA — Primary analysis:Group 2 vs 3. Key secondary analysis: Group 1 vs 3. Multiple comparisons for the analysis of the primary endpoint were controlled at the 5% level; Study baseline FEV1 as a covariate and treatment group as fixed effect

2. Secondary Outcome: Time-normalized Area From Study Baseline Curve for FEV1 Over 0-12 Hours (nAUC0-12B)
Time Frame: 0-12 hours following two weeks of dosing
Population: Total number of subjects in each arm: 76, 80, 78
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 71 | 75 | 72
Liters | 0.118 [0.070 to 0.167] | 0.130 [0.084 to 0.177] | 0.242 [0.195 to 0.290]
Statistical Analysis 1: Comparison: Arformoterol 15 Mcg Twice Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA; Study baseline FEV1 as a covariate and treatment group as a fixed effect
Statistical Analysis 2: Comparison: Tiotropium 18 Mcg Once Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p = 0.001, ANCOVA; Study baseline FEV1 as a covariate and treatment group as a fixed effect

3. Secondary Outcome: Time Normalized Area Under the Change From Study Baseline Curve for FEV1 Over 12-24 Hours (nAUC12-24B)
Time Frame: Following 2 weeks of dosing
Population: Total number of subjects in each arm: 76, 80, 78
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 63 | 67 | 71
Liters | 0.094 [0.036 to 0.151] | 0.054 [0.008 to 0.101] | 0.217 [0.169 to 0.264]
Statistical Analysis 1: Comparison: Arformoterol 15 Mcg Twice Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p = 0.001, ANCOVA; Study baseline FEV1 as a covariate and treatment group as a fixed effect
Statistical Analysis 2: Comparison: Tiotropium 18 Mcg Once Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA; Study baseline FEV1 as a covariate and treatment group as a fixed effect

4. Secondary Outcome: Change in FEV1 From Study Baseline to the 24-hour Timepoint (Trough)
Description: Trough FEV1 is defined as the measurement collected approximately 24 hours after the first in-clinic double-blind dose at Week 0. Change is calculated as Week 2 24 hour post first dose FEV1 - Week 0 pre-first dose FEV1.
Time Frame: Following 2 weeks of dosing
Population: Total number of subjects in each arm: 76, 80, 78
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 69 | 73 | 74
Liters | 0.086 [0.031 to 0.141] | 0.080 [0.032 to 0.129] | 0.154 [0.103 to 0.206]
Statistical Analysis 1: Comparison: Arformoterol 15 Mcg Twice Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p = 0.073, ANCOVA; Study baseline FEV1 as a covariate and treatment group as a fixed effect
Statistical Analysis 2: Comparison: Tiotropium 18 Mcg Once Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p = 0.050, ANCOVA; Study baseline FEV1 as a covariate and treatment group as a fixed effect

5. Secondary Outcome: Change in FEV1 From Study Baseline at Each Assessed Timepoint Post First Dose of Study Medication
Description: Baseline is FEV1 measurement collected prior to the first double-blind dose at week 0. Change defined as Week 0 FEV1 - Week 2 pre first dose FEV1.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 76 | 80 | 78
Liters
  Week 0: immediately post first dose; N=76, 78, 78 | 0.132 (0.155) | -0.20 (0.084) | 0.139 (0.151)
  Week 0: 30 minutes post first dose; N=75, 78, 76 | 0.163 (0.137) | 0.056 (0.093) | 0.183 (0.152)
  Week 0: 1 hour post first dose; N=75, 78, 77 | 0.182 (0.150) | 0.106 (0.141) | 0.189 (0.161)
  Week 0: 2 hours post first dose; N=76, 78, 77 | 0.193 (0.156) | 0.140 (0.148) | 0.239 (0.170)
  Week 0: 4 hours post first dose; N=75, 77, 77 | 0.155 (0.169) | 0.120 (0.169) | 0.223 (0.189)
  Week 0: 6 hours post first dose; N=72, 74, 77 | 0.128 (0.156) | 0.125 (0.188) | 0.214 (0.184)
  Week 0: 8 hours post first dose; N=70, 73, 77 | 0.102 (0.183) | 0.109 (0.208) | 0.194 (0.180)
  Week 0: 10 hours post first dose; N=69, 71, 76 | 0.101 (0.150) | 0.111 (0.184) | 0.190 (0.176)
  Week 0: 12 hours post first dose; N=69, 71, 75 | 0.044 (0.181) | 0.094 (0.196) | 0.199 (0.202)
  Week 2: immediately post first dose; N=71, 75, 74 | 0.154 (0.207) | 0.066 (0.184) | 0.240 (0.206)
  Week 2: 30 minutes post first dose; N=70, 74, 74 | 0.188 (0.222) | 0.126 (0.200) | 0.280 (0.216)
  Week 2: 1 hour post first dose; N=71, 75, 73 | 0.185 (0.222) | 0.163 (0.251) | 0.308 (0.232)
  Week 2: 2 hours post first dose; N=71, 73, 74 | 0.213 (0.226) | 0.195 (0.248) | 0.330 (0.228)
  Week 2: 4 hours post first dose; N=69, 72, 74 | 0.154 (0.227) | 0.164 (0.250) | 0.279 (0.239)
  Week 2: 6 hours post first dose; N=69, 72, 73 | 0.123 (0.211) | 0.143 (0.226) | 0.266 (0.208)
  Week 2: 8 hours post first dose; N=69, 70, 74 | 0.067 (0.221) | 0.138 (0.233) | 0.220 (0.215)
  Week 2: 10 hours post first dose; N=69, 71, 71 | 0.054 (0.224) | 0.109 (0.179) | 0.205 (0.211)
  Week 2: 12 hours post first dose; N=63, 67, 71 | 0.035 (0.211) | 0.101 (0.204) | 0.189 (0.210)
  Week 2: immediately post second dose; N=65, 67, 72 | 0.115 (0.223) | 0.040 (0.215) | 0.235 (0.202)
  Week 2: 12.5 hours post first dose; N=65, 66, 72 | 0.143 (0.235) | 0.063 (0.213) | 0.270 (0.214)
  Week 2: 13 hours post first dose; N=63, 68, 72 | 0.159 (0.234) | 0.061 (0.196) | 0.272 (0.220)
  Week 2: 14 hours post first dose; N=65, 71, 72 | 0.182 (0.248) | 0.068 (0.221) | 0.292 (0.234)
  Week 2: 16 hours post first dose; N=63, 70, 71 | 0.114 (0.233) | 0.048 (0.239) | 0.240 (0.216)
  Week 2: 23 hours post first dose; N=70, 74, 74 | 0.040 (0.236) | -0.006 (0.212) | 0.145 (0.208)
  Week 2: 24 hours post first dose; N=69, 73, 74 | 0.086 (0.229) | 0.080 (0.207) | 0.154 (0.223)

6. Secondary Outcome: Change in FEV1 Percent of Predicted From Study Baseline at Each Assessed Timepoint Post First Dose of Study Medication
Description: Baseline is FEV1 collected prior to first double-blind dose at week 0. Change is defined as Week 0 FEV1 percent predicted - Week 2 pre first dose FEV1 percent predicted.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Percent of predicted FEV1
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 76 | 80 | 78
Percent of predicted FEV1
  Week 0: Immediately post first dose; N=76, 78, 78 | 4.3 (4.6) | -0.6 (2.5) | 4.7 (4.9)
  Week 0: 30 minutes post first dose; N=75, 78, 76 | 5.5 (4.4) | 2.0 (3.2) | 6.1 (5.2)
  Week 0: 1 hour post first dose; N-75, 78, 77 | 6.1 (4.8) | 3.5 (4.6) | 6.3 (5.4)
  Week 0: 2 hours post first dose; N=76, 78, 77 | 6.6 (5.0) | 4.7 (5.1) | 8.1 (5.7)
  Week 0: 4 hours post first dose; N=75, 77, 77 | 5.3 (5.5) | 4.0 (5.3) | 7.5 (6.3)
  Week 0: 6 hours post first dose; N=72, 74, 77 | 4.4 (5.0) | 4.1 (5.9) | 7.3 (6.3)
  Week 0: 8 hours post first dose; N=70, 73, 77 | 3.5 (5.5) | 3.5 (6.5) | 6.6 (6.2)
  Week 0: 10 hours post first dose; N=69, 71, 76 | 3.3 (4.6) | 3.7 (5.6) | 6.5 (5.9)
  Week 0: 12 hours post first dose; N=69, 71, 75 | 1.6 (6.0) | 2.9 (6.1) | 6.7 (6.6)
  Week 2: Immediately post first dose; N=71, 75, 74 | 5.1 (6.4) | 1.9 (5.9) | 8.0 (6.7)
  Week 2: 30 minutes post first dose; N=70, 74, 74 | 6.2 (7.0) | 4.0 (6.3) | 9.3 (6.9)
  Week 2: 1 hour post first dose; N=71, 75, 73 | 6.2 (7.1) | 5.2 (7.6) | 10.2 (7.3)
  Week 2: 2 hours post first dose; N=71, 73, 74 | 7.1 (7.1) | 6.3 (7.3) | 11.0 (7.4)
  Week 2: 4 hours post first dose; N=69, 72, 74 | 5.1 (7.4) | 5.1 (7.5) | 9.2 (7.6)
  Week 2: 6 hours post first dose; N=69, 72, 73 | 4.0 (6.3) | 4.7 (6.9) | 8.8 (6.6)
  Week 2: 8 hours post first dose; N=69, 70, 74 | 2.0 (7.0) | 4.4 (7.1) | 7.4 (6.9)
  Week 2: 10 hours post first dose; N=69, 71, 71 | 1.8 (7.2) | 3.5 (5.7) | 6.8 (6.8)
  Week 2: 12 hours post first dose; N=63, 67, 71 | 1.3 (6.7) | 3.4 (6.3) | 6.3 (6.9)
  Week 2: Immediately post second dose; N=65, 67, 72 | 3.8 (6.9) | 1.1 (6.8) | 7.8 (6.6)
  Week 2: 12.5 hours post first dose; N=65, 66, 72 | 4.9 (7.2) | 2.0 (6.5) | 9.0 (7.0)
  Week 2: 13 hours post first dose; N=63, 68, 72 | 5.4 (7.3) | 1.8 (6.0) | 9.1 (7.1)
  Week 2: 14 hours post first dose; N=65, 71, 72 | 6.0 (7.6) | 2.0 (6.7) | 9.8 (7.7)
  Week 2: 16 hours post first dose; N=63, 70, 71 | 3.9 (7.1) | 1.4 (7.3) | 8.0 (6.9)
  Week 2: 23 hours post first dose; N=70, 74, 74 | 1.3 (7.0) | -0.2 (6.5) | 4.8 (6.7)
  Week 2: 24 hours post first dose; N=69, 73, 74 | 2.8 (6.9) | 2.6 (6.6) | 5.2 (7.2)

7. Secondary Outcome: Peak Change in FEV1 Over 12 Hours Post Dose From Study Baseline
Description: 12 hour peak change in FEV1 is defined as maximum of the post dose changes through the nominal 12 hour assessment.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 76 | 80 | 78
Liters
  Week 0; N=76, 79, 78 | 0.264 [0.231 to 0.296] | 0.218 [0.179 to 0.257] | 0.311 [0.272 to 0.350]
  Week 2; N=71, 75, 74 | 0.273 [0.223 to 0.324] | 0.265 [0.212 to 0.319] | 0.379 [0.328 to 0.430]
Statistical Analysis 1: Comparison: Arformoterol 15 Mcg Twice Daily vs Arformoterol /Tiotropium; Week 0 comparisons; Test type: Superiority or Other; p = 0.060, ANCOVA; Week 0 comparisons: Study baseline FEV1 as a covariate and treatment group as a fixed effect
Statistical Analysis 2: Comparison: Tiotropium 18 Mcg Once Daily vs Arformoterol /Tiotropium; Week 0; Test type: Superiority or Other; p < 0.001, ANCOVA; Study baseline FEV1 as a covariate and treatment group as a fixed effect
Statistical Analysis 3: Comparison: Arformoterol 15 Mcg Twice Daily vs Arformoterol /Tiotropium; Week 2 comparisons; Test type: Superiority or Other; p = 0.004, ANCOVA; Week 2 comparisons: Study baseline FEV1 as a covariate and treatment group as a fixed effect
Statistical Analysis 4: Comparison: Tiotropium 18 Mcg Once Daily vs Arformoterol /Tiotropium; Week 2 comparisons; Test type: Superiority or Other; p = 0.002, ANCOVA; Week 2 comparisons: Study baseline FEV1 as a covariate and treatment group as a fixed effect

8. Secondary Outcome: Time to Onset in Participants Who Achieved a 10% Increase in FEV1 From Visit Predose After 2 Weeks
Description: Analyzed from end of dosing to 12 hours.
Time Frame: 2 weeks
Population: Total number of subjects in each arm: 76, 80, 78.
Measure: Median (Full Range); unit: Hours
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 42 | 45 | 48
Hours | 0.39 [0.02 to 7.03] | 0.72 [0.02 to 10.07] | 0.17 [0.03 to 6.80]

9. Secondary Outcome: Time to Onset in Participants Who Achieved a 15% Increase in FEV1 From Visit Predose After 2 Weeks
Description: Analyzed from end of dosing to 12 hours.
Time Frame: 2 weeks
Population: Total number of subjects in each arm: 76, 80, 78.
Measure: Median (Full Range); unit: Hours
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 30 | 32 | 34
Hours | 0.76 [0.02 to 7.90] | 1.29 [0.03 to 7.25] | 0.39 [0.08 to 10.88]

10. Secondary Outcome: Change in Inspiratory Capacity From Study Baseline to the 24 Hour Timepoint (Trough) Following 2 Weeks of Dosing
Description: Trough Inspiratory Capacity is defined as the measurement collected approximately 24 hours after the first in clinic double-blind treatment dose at week 0. Change is calculated as Week 2 24 hr post dose IC - Week 0 pre first dose IC.
Time Frame: 2 weeks
Population: Total number of subjects in each arm: 76, 80, 78
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 66 | 69 | 70
Liters | 0.074 [0.00 to 0.147] | 0.023 [-0.047 to 0.094] | 0.150 [0.065 to 0.235]
Statistical Analysis 1: Comparison: Arformoterol 15 Mcg Twice Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p = 0.206, ANCOVA; Study baseline Inspiratory Capacity as a covariate and treatment group as a fixed effect
Statistical Analysis 2: Comparison: Tiotropium 18 Mcg Once Daily vs Arformoterol /Tiotropium; Test type: Superiority or Other; p = 0.025, ANCOVA; Study baseline Inspiratory Capacity as a covariate and treatment group as a fixed effect

11. Secondary Outcome: Change in Forced Vital Capacity (FVC) From Study Baseline at Each Assessed Post Dose Timepoint
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 76 | 80 | 78
Liters
  Week 0: Immediately post first dose; N=76, 78, 78 | 0.276 (0.270) | -0.031 (0.165) | 0.259 (0.305)
  Week 0: 30 minutes post first dose; N=75, 78, 76 | 0.312 (0.267) | 0.122 (0.210) | 0.323 (0.347)
  Week 0: 1 hour post first dose; N=75, 78, 77 | 0.344 (0.275) | 0.197 (0.283) | 0.351 (0.348)
  Week 0: 2 hours post first dose; N=76, 78, 77 | 0.376 (0.319) | 0.248 (0.279) | 0.429 (0.366)
  Week 0: 4 hours post first dose; N=75, 77, 77 | 0.291 (0.341) | 0.206 (0.293) | 0.392 (0.375)
  Week 0: 6 hours post first dose; N=72, 74, 77 | 0.242 (0.303) | 0.195 (0.327) | 0.371 (0.352)
  Week 0: 8 hours post first dose; N=70, 73, 77 | 0.207 (0.334) | 0.159 (0.360) | 0.338 (0.325)
  Week 0: 10 hours post first dose; N=69, 71, 76 | 0.209 (0.267) | 0.175 (0.311) | 0.346 (0.357)
  Week 0: 12 hours post first dose; N=69, 71, 75 | 0.131 (0.299) | 0.146 (0.325) | 0.344 (0.352)
  Week 2: Immediately post first dose; N=71, 75, 74 | 0.293 (0.368) | 0.055 (0.301) | 0.389 (0.392)
  Week 2: 30 minutes post first dose; N=70, 74, 74 | 0.343 (0.381) | 0.203 (0.350) | 0.461 (0.425)
  Week 2: 1 hour post first dose; N=71, 75, 73 | 0.350 (0.397) | 0.224 (0.408) | 0.487 (0.426)
  Week 2: 2 hours post first dose; N=71, 73, 74 | 0.380 (0.389) | 0.290 (0.387) | 0.526 (0.426)
  Week 2: 4 hours post first dose; N=69, 72, 74 | 0.265 (0.342) | 0.221 (0.372) | 0.461 (0.441)
  Week 2: 6 hours post first dose; N=69, 72, 73 | 0.202 (0.322) | 0.209 (0.356) | 0.413 (0.383)
  Week 2: 8 hours post first dose; N=69, 70, 74 | 0.136 (0.347) | 0.214 (0.319) | 0.349 (0.387)
  Week 2: 10 hours post first dose; N=69, 71, 71 | 0.098 (0.364) | 0.158 (0.278) | 0.323 (0.379)
  Week 2: 12 hours post first dose; N=63, 67, 71 | 0.087 (0.340) | 0.124 (0.365) | 0.301 (0.398)
  Week 2: Immediately post second dose; N=65, 67, 72 | 0.210 (0.397) | 0.034 (0.356) | 0.360 (0.385)
  Week 2: 12.5 hours post first dose; N=65, 66, 72 | 0.262 (0.416) | 0.087 (0.359) | 0.399 (0.407)
  Week 2: 13 hours post first dose; N=63, 68, 72 | 0.307 (0.376) | 0.082 (0.329) | 0.424 (0.432)
  Week 2: 14 hours post first dose; N=65, 71, 72 | 0.343 (0.386) | 0.110 (0.342) | 0.459 (0.445)
  Week 2: 16 hours post first dose; N=63, 70, 71 | 0.215 (0.374) | 0.098 (0.361) | 0.374 (0.422)
  Week 2: 23 hours post first dose; N=70, 74, 74 | 0.082 (0.363) | -0.011 (0.340) | 0.226 (0.345)
  Week 2: 24 hours post first dose; N=69, 73, 74 | 0.138 (0.365) | 0.115 (0.335) | 0.250 (0.408)

12. Secondary Outcome: Levalbuterol Metered Dose Inhaler (MDI) (Rescue Medication) Use in Days Per Week
Description: Overall: Average of the levalbuterol usage in days per week over the 2 week period. Mean number of days/week=number of days levalbuterol used during time period, divided by number of days in the period, multiplied by 7. An actuation is one puff of levalbuterol.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: Days per week
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 76 | 80 | 78
Days per week
  Baseline: Number of days used per week | 4.44 [3.79 to 5.08] | 4.27 [3.61 to 4.92] | 4.57 [3.94 to 5.20]
  Overall: Number of days used per week | 2.16 [1.57 to 2.75] | 1.94 [1.40 to 2.47] | 1.38 [0.87 to 1.89]

13. Secondary Outcome: Levalbuterol Metered Dose Inhaler (MDI) Rescue Medication Use in Actuations Per Day
Description: Overall: Average of the usage in number of actuations per day over the 2 week period. An actuation is one puff of levalbuterol. Mean number of actuations/day=number actuations used during time period, divided by number of days in time period.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: Actuations per day
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 76 | 80 | 78
Actuations per day
  Baseline: Number of actuations per day | 3.24 [2.50 to 3.98] | 2.77 [2.16 to 3.39] | 3.08 [2.47 to 3.69]
  Overall: Number of actuations per day | 1.18 [0.75 to 1.61] | 1.00 [0.59 to 1.40] | 0.68 [0.36 to 1.00]

14. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score
Description: TDI Focal score (range -9 to 9) is defined as the sum of function impairment, magnitude of task, and magnitude of effort (each on a -3 to 3 scale). A score of -9 is maximum worsening and 9 is maximum improvement.
Time Frame: 2 weeks
Population: Total number of subjects in each arm: 76, 80, 78
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 75 | 77 | 77
Units on a scale | 2.28 (2.39) | 1.79 (2.83) | 3.13 (2.44)

15. Secondary Outcome: Number of Participants With a >= 1 Unit of Improvement in the TDI Focal Score
Description: A Greater than or Equal to 1 unit of Improvement in the TDI Focal Score is considered to be clinically important.
Time Frame: 2 weeks
Population: Total number of subjects in each arm: 76, 80, 78
Measure: Number; unit: Participants
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 75 | 77 | 77
Participants | 50 | 44 | 60

16. Secondary Outcome: Percentage of Participants With a >=1 Unit Improvement in Transition Dysnea Index (TDI) Focal Score
Description: A Greater than or Equal to 1 unit of Improvement in the TDI Focal Score is considered to be clinically important.
Time Frame: 2 weeks
Population: Total number of subjects in each arm: 76, 80, 78
Measure: Number; unit: Percentage of participants
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Number analyzed (Participants) | 75 | 77 | 77
Percentage of participants | 66.67 | 57.14 | 77.92

ADVERSE EVENTS:
Arm/Group | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Serious Adverse Events (participants affected / at risk) | 1 | 0 | 0
Other Adverse Events (participants affected / at risk) | 8 | 12 | 16
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Small Intestinal Obstruction (Gastrointestinal disorders) | 1/76 (1) | 0/80 (0) | 0/78 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Arformoterol 15 Mcg Twice Daily | Tiotropium 18 Mcg Once Daily | Arformoterol /Tiotropium
Diarrhoea (Gastrointestinal disorders) | 0/76 (0) | 0/80 (0) | 2/78 (2)
Nausea (Gastrointestinal disorders) | 1/76 (2) | 2/80 (2) | 0/78 (0)
Chest Pain (General disorders) | 0/76 (0) | 0/80 (0) | 2/78 (2)
Bronchitis (Infections and infestations) | 2/76 (2) | 0/80 (0) | 0/78 (0)
Dizziness (Nervous system disorders) | 1/76 (1) | 1/80 (1) | 2/78 (2)
Headache (Nervous system disorders) | 1/76 (2) | 3/80 (4) | 4/78 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/76 (1) | 2/80 (2) | 2/78 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0/76 (0) | 2/80 (2) | 0/78 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2/76 (3) | 1/80 (1) | 2/78 (2)
Hypertension (Vascular disorders) | 0/76 (0) | 2/80 (2) | 2/78 (2)

LIMITATIONS AND CAVEATS:
As of October 24, 2008, Sepracor is unaware of any limitations or caveats associated with this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.